CLINICAL TRIAL: NCT00828035
Title: Light Endoscopic Robot Use in Abdominal and Urological Laparoscopic Surgery
Brief Title: Light Endoscopic Robot Use in Laparoscopic Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Principal Investigator, AdministrateurCIC, principal investigator, University Hospital, Grenoble
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DCIC 03 39; ENDOCONTROL company
Record Dates: First submitted 2009-01-22; First posted 2009-01-23 (Estimated); Last update posted 2012-09-18 (Estimated); Status verified 2012-09

CONDITIONS: Laparoscopy
Keywords: robotics; laparoscopy; surgery; computer assisted
MeSH Terms: interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1, REL (Other): rel group : patients with light endoscopic robot
  Interventions: Procedure: laparoscopic surgery
- 2, AO (Active Comparator): AO group : Patients with surgery assistant
  Interventions: Procedure: laparoscopic surgery

INTERVENTIONS:
Procedure: laparoscopic surgery — comparison of two different laparoscopic surgeries : robot versus human
  Other Names: robotic laparoscopic surgery; robotic abdominal laparoscopic surgery; robotic urological laparoscopic surgery

SUMMARY:
Light Endoscopic Robot evaluation in abdominal and urological laparoscopic surgery : surgery with surgeon and robot (REL group = new treatment) versus surgery with surgeon and assistant (AO group - standard treatment)

Primary outcome measure : Number of useful hands (light endoscopic robot = one useful mechanical hand)

ELIGIBILITY:
Inclusion Criteria:

* Laparoscopic surgery indicated
* Subject with ASA Score 1, 2 or 3
* Subject with health and social protection
* 18 years of age or older
* Written Informed Consent

Exclusion Criteria:

* Subject is pregnant or lactating
* Subject in jail
* Subject hospitalizes without consent
* Protected persons aged 18 years or older
* Subject participated in another study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-04; Primary Completion 2008-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
Number of useful hands, robot as a useful mechanical hand | one month

SECONDARY OUTCOMES:
To evaluate reliability and limits of light endoscopic robot : Number of breakdown, failure (manipulation, voice recognition, other ) | one month
Compare surgeon's visual comfort in two groups (REL group and AO group) : evaluate scale of surgeon's visual comfort during surgery | one month
Compare surgery's periods | one month
Evaluate complications : Number of complications (per operative, post operative) | one month
Evaluate medical and paramedical use of light endoscopic robot : apprentice time, labour time | one month
Medical and economic evaluation : cost benefit analysis : human cost, cost | one month

CONTACTS AND LOCATIONS:
Overall Officials: Christian LETOUBLON, MD, Principal Investigator — University Hospital, Grenoble; Jean-Jacques RAMBEAUD, MD, Principal Investigator — University Hospital, Grenoble
Locations (2):
- France (2):
  - University Hospital, Grenoble, Grenoble, Isère
  - University Hospital, Saint-Etienne, Saint-Étienne-de-Montluc, Pays de la Loire Region

REFERENCES:
- [Background] Long JA, Descotes JL, Skowron O, Troccaz J, Cinquin P, Boillot B, Terrier N, Rambeaud JJ. [Use of robotics in laparoscopic urological surgery: state of the art]. Prog Urol. 2006 Feb;16(1):3-11. French. PMID 16526532
- [Background] Aiono S, Gilbert JM, Soin B, Finlay PA, Gordan A. Controlled trial of the introduction of a robotic camera assistant (EndoAssist) for laparoscopic cholecystectomy. Surg Endosc. 2002 Sep;16(9):1267-70. doi: 10.1007/s00464-001-9174-7. Epub 2002 Jun 14. PMID 12235507
- [Derived] Jarry J, Moreau Gaudry A, Long JA, Chipon E, Cinquin P, Faucheron JL. Miniaturized robotic laparoscope-holder for rectopexy: first results of a prospective study. J Laparoendosc Adv Surg Tech A. 2013 Apr;23(4):351-5. doi: 10.1089/lap.2012.0233. Epub 2013 Mar 11. PMID 23477369